CLINICAL TRIAL: NCT04578496
Title: A Phase III, Safety Extension Study in Patients With Erythropoietic Protoporphyria (EPP)
Brief Title: A Safety Extension Study in Patients With Erythropoietic Protoporphyria (EPP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUV037
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Erythropoietic Protoporphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — afamelanotide

ARMS (1):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide

SUMMARY:
The main objectives of the study were to evaluate the safety and tolerability of afamelanotide by measuring treatment emergent adverse events (AEs) and to determine whether afamelanotide can improve the quality of life of EPP patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects with a positive diagnosis of EPP who successfully completed the CUV017 or CUV029 studies;
* aged 18-75 years (inclusive);
* provide written informed patient consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* any serious adverse event considered to be related to afamelanotide or the polymer contained in the implant;
* any allergy to lignocaine or other local anaesthetic to be used during the administration of the study medication;
* EPP patients with significant hepatic involvement;
* personal history of melanoma or dysplastic nevus syndrome;
* current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions;
* any evidence of clinically significant organ dysfunction or any clinically significant deviation from normal in the clinical or laboratory determinations;
* acute history of drug or alcohol abuse (in the last 12 months);
* female who is pregnant (confirmed by positive serum β-Human Chorionic Gonadotropin (HCG) pregnancy test prior to baseline) or lactating;
* females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device);
* sexually active men with partners of child-bearing potential not using barrier contraception during the trial and for a period of three months thereafter;
* participation in a clinical trial for an investigational agent within 30 days prior to the screening visit;
* prior and concomitant therapy with medications which may interfere with the objectives of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Bilbao, Study Director — Clinuvel Pharmaceuticals Limited

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Afamelanotide
Started | 16
Completed | 12
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Afamelanotide
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Measured Using the EPP-quality of Life Questionnaire (EPP-QoL).
Description: The EPP-QoL is presented as 15 questions aiming at measuring how the condition has affected the patient over the last 2 months. Each question is answered on a categorical scale. The maximum score is calculated by summing the score of each question resulting in a maximum of 100 and a minimum of 0. The higher the score, the better the quality of life.
Time Frame: Baseline, Day 60, Day 120, Day 180 or early termination (ET) (if applicable)
Population: Intent-to-treat population
Measure: Median (Full Range); unit: EPP-QoL score
Arm/Group | Afamelanotide
Number analyzed (Participants) | 13
EPP-QoL score
  Day 60 | 27.8 [-56 to 75]
  Day 120 | 59.7 [11 to 85]
  Day 180 or ET | 56.9 [8 to 67]

2. Primary Outcome: Change in Quality of Life Measured Using the Dermatology Life Quality Index Questionnaire (DLQI)
Description: The DLQI questionnaire consists of 10 questions, each answered on a categorical scale. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline, Day 60, Day 120, Day 180 or early termination (ET) (if applicable)
Population: Intent-to-treat population
Measure: Median (Full Range); unit: DLQI score
Arm/Group | Afamelanotide
Number analyzed (Participants) | 13
DLQI score
  Day 60 | -5 [-17 to 1]
  Day 120 | -4.5 [-17 to 0]
  Day 180 or ET | -5 [-17 to 0]

ADVERSE EVENTS:
Description: The adverse event reported below is an adverse event assessed to be related to the study drug by the investigator.
Arm/Group | Afamelanotide
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afamelanotide (N=16)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No